CLINICAL TRIAL: NCT07036666
Title: An Open Label Study Assessing the Impact of a Women's Health Formulation on Vaginal Health and the Microbial Community
Brief Title: A Study Assessing the Impact of a Women's Health Formulation on Vaginal Health and the Microbial Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RADX-C003-N
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-06

CONDITIONS: Women's Health

STUDY DESIGN:
Intervention Model Description: Single arm, 5-week (4 week product consumption), open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Product (Experimental): Women's (vaginal) health active product
  Interventions: Dietary Supplement: Active Product

INTERVENTIONS:
Dietary Supplement: Active Product — Women's (vaginal) Health Active Product

SUMMARY:
An open label study assessing the impact of a women's health formulation on vaginal health and the microbial community

DETAILED DESCRIPTION:
This is an open label study conducted with adult participants, assigned female at birth, residing in the United States.

Eligible participants will (1) endorse a desire for better vaginal health and (2) have the opportunity for meaningful improvement (at least 30%) in their primary health outcome.

Participants that report a known cardiac dysfunction, liver or kidney disease may be excluded. Participants that report a known contraindication or with well-established, significant safety concerns due to illness will be excluded. Heavy drinkers and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Participants that report taking medications with a known contraindication or with well-established, significant safety concerns will be excluded.

Self-reported data are collected electronically from eligible participants over 5 weeks. Participant reports of health indicators will be collected at baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all the following criteria:

  * Adults, assigned female at birth, 21-65 years of age at the time of electronic consent, inclusive of all ethnicities, races
  * Resides in the United States
  * Endorses better vaginal health as a primary desire
  * Has the opportunity for at least 30% improvement in their primary health outcome (i.e., Vaginal Health Survey score ≥ 14 at screening)
  * Willingness to complete a vaginal biospecimen at 2 timepoints

Exclusion Criteria:

* Individuals who report any of the following during screening will be excluded from participation:

  * Report being pregnant, trying to become pregnant, or breastfeeding
  * Unable to provide a valid US shipping address and mobile phone number ● Reports current enrollment in another clinical trial
  * Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
  * Unable to read and understand English
  * Reports a current and/or recent (up to 3 months ago) major illness and/or surgery that poses a known, significant safety risk.
  * Reports a diagnosis of cardiac dysfunction, liver or kidney disease that presents a known contraindication and/or a significant safety risk with any of the study product ingredients.

    o NYHA Class III or IV congestive heart failure, atrial fibrillation, uncontrolled arrhythmias, cirrhosis, end-stage liver disease, stage 3b or 4 chronic kidney disease, or kidney failure
  * Reports taking medications that have a well-established moderate or severe interaction, posing a substantial safety risk with any of the study product ingredients. o Anticoagulants, antihypertensives, anxiolytics, antidepressants, chemotherapy, immunotherapy, sedative hypnotics, seizure medications, medications that warn against grapefruit consumption, corticosteroids at doses greater than 5 mg per day, diabetic medications, oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection, antipsychotics, MAOIs, or thyroid products
  * Reports current use of the primary ingredient(s) and/or similar product(s) to the active study product(s) that may limit the effects of the study products
  * Participants must not be undergoing treatment for bacterial vaginosis (ABX) - they will be ineligible if they answer yes to antimicrobials
  * Participants must not be using prescription or over- the- counter (OTC) treatments for bacterial vaginosis or yeast infections
  * Participants must not be have been diagnosed with a urinary tract infection (UTI) in the past 3 months
  * Lack of reliable daily access to the internet

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Change in Vaginal Health | 5 weeks
  Difference between rates of change over time in vaginal health score as assessed by Vaginal Health Survey (scale 6-30; where the higher scores correspond to worse vaginal health)

SECONDARY OUTCOMES:
Change in Digestion-related Quality of Life (DQLQ) | 5 weeks
  Difference between rates of change over time in DQLQ score as assessed by Digestion-related Quality of Life survey (scale 0-9; where the higher scores correspond to worse GI-related quality of life)
Change in Overall Health Profile | 5 weeks
  Difference between rates of change over time in overall health score as assessed by Patient Reported Outcome Measurement System (PROMIS) 29+2 Profile (PROPr consists of 7 health domains: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognitive function abilities; PROPr t-score score range = -.022 to 1; higher scores indicate greater overall health)
Minimal Clinical Importance Difference (MCID) in Vaginal Health | 5 weeks
  Likelihood of achieving a MCID in vaginal health, as measured by Vaginal Health Survey (scale 6-30; where the higher scores correspond to worse vaginal health)
Minimal Clinical Importance Difference (MCID) in Digestion-related Quality of Life (DQLQ) | 5 weeks
  Likelihood of achieving a MCID in overall health, as measured by Digestion-related Quality of Life survey (scale 0-9; where the higher scores correspond to worse GI-related quality of life)
Minimal Clinical Importance Difference (MCID) in Overall Health Profile | 5 weeks
  Likelihood of achieving a MCID in digestion-related quality of life, as measured by (PROMIS) 29+2 Profile (PROPr consists of 7 health domains: physical function, anxiety, depression, fatigue, sleep disturbance, ability to participate in social roles and activities, pain interference, cognitive function abilities; PROPr t-score score range = -.022 to 1; higher scores indicate greater overall health)
Vaginal Total Lactobacilli Abundance | 5 weeks
  Estimate the mean change in biomarker levels from baseline
Vaginal Community State Type (CST) | 5 weeks
  Estimate the mean change in biomarker levels from baseline
Vaginal pH | 5 weeks
  Estimate the mean change in biomarker levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Susan Hewlings, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside Radicle Science collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com